CLINICAL TRIAL: NCT00299858
Title: Effect of Theophylline on Exercise Capacity and Lung Function in COPD Patients Receiving Long-acting Inhaled Bronchodilator Therapy
Brief Title: Theophylline in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ontario Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006036-01H
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: COPD
Keywords: Chronic Obstructive Pulmonary Disease; Theophylline; Exercise testing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Theophylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group (Active Comparator): Patients will be given theophylline, titrated to optimal blood levels, for a period of 4 weeks.
  Interventions: Drug: Theophylline
- Placebo group (Placebo Comparator): Patients will receive placebo pills for a period of 4 weeks.
  Interventions: Drug: Theophylline

INTERVENTIONS:
Drug: Theophylline — Patients assigned to study group, will receive slow-release theophylline at a dose of 10 mg/kg, titrated to blood levels between 55-110 umol/L, for a period of 4 weeks.
  Patients assigned to placebo group will receive identical-appearing placebo tablets for the same period of time.

SUMMARY:
This will be a prospective randomized double-blinded parallel group clinical trial evaluating the short-term effects of theophylline therapy on exercise duration and lung function in patients with chronic obstructive pulmonary disease already receiving both tiotropium and a long-acting beta-agonist (salmeterol or formoterol).

DETAILED DESCRIPTION:
Objective:

The primary objectives of this study is to assess the effects of 4 weeks of theophylline therapy on exercise performance and lung function in patients with COPD already receiving combination inhaled long-acting bronchodilator therapy.

Background:

The latest Canadian COPD guidelines recommend the use of long-acting bronchodilators in patients who continue to experience symptoms despite as-needed use of short-acting bronchodilators. Unfortunately, patients with severe COPD may continue to experience symptoms despite use of both long-acting beta-agonists and anticholinergics. For these patients, the Canadian guidelines recommend a trial of theophylline. Studies have shown that theophylline can reduce symptoms and improve exercise performance, however, the use of theophylline is limited by its narrow therapeutic window and multiple drug interactions. Despite recommendations, it remains unknown whether theophylline provides any additional benefit for COPD patients already receiving combined long-acting bronchodilator therapy. No study has evaluated the effect of theophylline in patients already receiving both long-acting beta-agonist and long-acting anticholinergic therapy.

Methods:

This will be a prospective randomized double-blinded parallel group clinical trial evaluating the short-term effects of theophylline therapy on exercise duration and lung function in patients already receiving both tiotropium and a long-acting beta-agonist (salmeterol or formoterol). Twenty-four patients with moderate to severe COPD who are already using tiotropium and long-acting beta agonists will be randomized to receive either: a) 4 weeks of oral theophylline dosed to achieve therapeutic blood levels, or b) 4 weeks of identical placebo therapy. Only patients with stable COPD (no exacerbations nor changes in medications over the last 2 months) and no contraindications to exercise testing or theophylline use will be enrolled. All patients will undergo baseline pulmonary function testing and incremental and constant load exercise testing prior to randomization. PFTs and constant load exercise testing will be repeated after 4 weeks of therapy. Patients will be instructed to report adverse events and will have their theophylline dose adjusted to ensure therapeutic bloods levels (55-110 umol/L), prior to repeat testing.

Outcome Measurements:

The primary outcome of interest will be the effect of theophylline on exercise duration during constant load (75% maximum) exercise testing. The study will be powered to detect a 20% greater improvement in exercise duration for the theophylline-treated group. Secondary outcome measures will include changes in spirometry (FEV1) and lung volumes.

Anticipated results:

Exercise duration (on constant load exercise testing) was chosen as the primary endpoint of this study because it has been shown to be a reproducible and highly responsive measure for physiologic benefit in COPD. It is unknown whether theophylline will provide any additional increase in exercise duration, when added to a combined long-acting bronchodilator regimen. If an improvement is found with theophylline, a follow-up study of larger size and longer duration will be required to investigate whether this benefit will translate into improvements in clinical outcomes such as quality of life or frequency of exacerbations. Alternatively, if no improvement can be detected, the current COPD treatment recommendation should be re-evaluated.

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosis of COPD, that is at least "moderate" in severity according to GOLD guidelines (FEV1 60% predicted and FEV1/FVC ratio 70%).

clinically stable (no exacerbations nor changes in medications over the previous two months.

taking tiotropium 18ug qd and either salmeterol 50ug bid or formoterol 12 ug bid (the use of inhaled corticosteroids is not required but is permitted as long as there have been no dose changes over the last 2 months).

Exclusion Criteria:

Lung disease other than COPD (e.g: asthma, interstitial lung disease)

Non-pulmonary comorbidity that may potentially limit exercise capacity (e.g: cardiac disease, arthritis) or be exacerbated by theophylline use.

History of adverse response to theophylline or condition that may increase likelihood of adverse reaction with theophylline (cardiac disease, liver disease, renal impairment, thyroid disease)

Use of theophylline over last two months.

Use of a medication that may potentially interact with theophylline (e.g. warfarin, digoxin)

Patients currently enrolled (or scheduled to be enrolled) in a pulmonary rehabilitation program will not be accepted until after completion of the program (as this may potentially affect exercise performance).

Use of systemic corticosteroid therapy (this may affect peripheral muscle function)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Exercise duration during constant load (75% maximum) exercise testing | End of 4 week treatment period

SECONDARY OUTCOMES:
Changes in spirometry (FEV1) Changes in lung volumes | End of 4 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Nha Voduc, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital, General campus, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Voduc N, Alvarez GG, Amjadi K, Tessier C, Sabri E, Aaron SD. Effect of theophylline on exercise capacity in COPD patients treated with combination long-acting bronchodilator therapy: a pilot study. Int J Chron Obstruct Pulmon Dis. 2012;7:245-52. doi: 10.2147/COPD.S29990. Epub 2012 Mar 29. PMID 22563244